CLINICAL TRIAL: NCT02946723
Title: A Study to Compare the Efficacy and Safety of Ultrasound Guided Lead Implantation for Sacral Neuromodulation (SNM) in Subjects With Overactive Bladder (OAB)With X-Ray Guided Technique
Brief Title: A Study to Compare the Efficacy and Safety of Ultrasound Guided Lead Implantation for Sacral Neuromodulation (SNM) in Subjects With Overactive Bladder (OAB) With X-Ray Guided Technique
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Pins Medical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PINS-022
Record Dates: First submitted 2016-10-25; First posted 2016-10-27 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Refractory Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — High-Energy Shock Waves; X-Rays

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- US group (Experimental): lead implantation surgery for SNM using ultrasound guided technique
  Interventions: Procedure: ultrasound
- X-ray group (Sham Comparator): lead implantation surgery for SNM using X-ray guided technique
  Interventions: Procedure: X-ray

INTERVENTIONS:
Procedure: ultrasound — Lead implantation surgery for SNM using ultrasound guided technique
  Arms: US group
Procedure: X-ray — Lead implantation surgery for SNM using X-ray technique
  Arms: X-ray group

SUMMARY:
Overactive bladder(OAB,Urgency) was determined by International Continence Society as Urinary urgency, usually accompanied by frequency and nocturia, with or without urgency urinary incontinence, in the absence of urinary tract infection (UTI) or other obvious pathology.The SNM treatment involves a two-stage surgical procedure performed under local anesthesia. The device include IPG (implantable programme generator) and lead. In the initial test phase, 1st stage, electrode is placed near the sacral nerve and requires a 2 weeks assessment. This allows your doctors and you to assess your initial response according to your voiding dairy and satisfaction. In 2nd stage, SNM procedure is implantation of the IPG.

X ray guidance is harmful to both patients and doctors, while ultrasound guidance is real time visual guidance ,easy to operate by doctors and a radiation free option to challenge anatomy. Urologists are skilled in both ultrasound operations and anatomy basics and dedicating to developing better guidance technique in surgery.

The study here compare the efficacy and safety of ultrasound versus X ray guidance technique in SNM.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 16 years;
2. Subjects suitable for SNM surgery;
3. Normal upper urinary tract function;
4. Bladder volume > 100 mL;
5. Good compliance and able to complete the follow-up assessments.

Exclusion Criteria:

1. Psychiatric or neurologic disabilities on neurologic evaluation such as multiple sclerosis, spinal cord injury, epilepsy, Parkinson's disease, stroke;
2. Bladder lithiasis or tumor (cystoscopy or ultrasonography);
3. Stress urinary incontinence;
4. Bladder outlet obstruction;
5. Diuresis > 3 liters per 24 hours;
6. Negative at the test period or previous treatment with SNM;
7. Pregnancy and plan to be pregnancy in 2 years.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-02; Primary Completion 2018-08 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Successful rate | 6 months post -IPG implantation
  Successful rate is the percentage of patients who experienced a successful result (≥50% improvements in baseline symptoms ) as recorded in voiding dairies.

SECONDARY OUTCOMES:
Adverse effect | During operation, 2 weeks post-lead implantation, 3 and 6 months post -IPG implantation
Guidance technique performance time | From beginning operation until successful lead placement is completed
Times of X-ray radiation | During operation
Overactive bladder symptom score (OABSS) | pre-operation baseline, 2 weeks post-lead implantation, 3 and 6 months post -IPG implantation
Quality of Life (QoL) scores | pre-operation baseline, 2 weeks post-lead implantation, 3 and 6 months post -IPG implantation